CLINICAL TRIAL: NCT03589274
Title: Testing CBT Models and Change Mechanisms for Alcohol Dependent Women
Acronym: WTPIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Elizabeth Epstein, Ph.D., Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-346R08x
Record Dates: First submitted 2018-06-08; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol use disorder; women; female specific therapy; cognitive behavior therapy; group therapy
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-FS-CBT (Experimental): In I-FS-CBT each participant saw a therapist weekly. The first session was 90 minutes long, and subsequent sessions were 60 minutes long. The I-FS-CBT manual included core CBT, motivational enhancement, and relapse prevention components. Two core thematic women's issues were integrated into each session via discussion and illustrative material: (a) self-confidence, and (b) self-care.
  Interventions: Behavioral: I-FS-CBT
- G-FS-CBT (Experimental): The G-FS-CBT manual included core CBT, motivational enhancement, and relapse prevention components. Two core thematic women's issues were integrated into each session via discussion and illustrative material: (a) self-confidence, and (b) self-care. The session organization was modified for a closed group format. The group treatment was designed to provide didactic presentation of coping skills and motivational enhancement material, and group discussion and rehearsal of new skills within a supportive atmosphere that facilitated mutual emotional support and support for abstinence.
  Interventions: Behavioral: G-FS-CBT

INTERVENTIONS:
Behavioral: I-FS-CBT — 12 manual-guided sessions of I-FS-CBT
  Arms: I-FS-CBT
Behavioral: G-FS-CBT — 12 manual-guided sessions of G-FS-CBT
  Arms: G-FS-CBT

SUMMARY:
The study has 4 specific aims: (1) To modify our existing Individual Female Specific Cognitive Behavioral Therapy (I-FS-CBT) for Alcohol Use Disorder (AUD) approach to treat women with alcohol dependence in a group format, Group Female Specific Cognitive Behavioral Therapy (G-FS-CBT); (2) To test the relative efficacy of I-FS-CBT and G-FS-CBT; (3) To test hypothesized mechanisms of change in drinking that are common to both treatments, including (a) coping skills and enhanced self-efficacy for abstinence; (b) enhanced sense of autonomy; (c) alleviation of negative affect, and (d) increased social network support for abstinence, and (4) To assess the relative cost-effectiveness of the individual and group treatment.

DETAILED DESCRIPTION:
Participants completed a telephone screen for initial eligibility and were scheduled for an in-person clinical intake interview. Consented women were scheduled for a baseline research interview (BL) approximately one week later. At the end of the BL, participants were randomized to treatment condition. During the 12 session treatment period, women completed assessments at the beginning and end of each therapy session on secondary outcome and therapy process variables.

In I-FS-CBT each participant saw a therapist weekly. The first session was 90 minutes long, and subsequent sessions were 60 minutes long. The I-FS-CBT manual included core CBT, motivational enhancement, and relapse prevention components. Two core thematic women's issues were integrated into each session via discussion and illustrative material: (a) self-confidence and (b) self-care.

The G-FS-CBT manual included material identical to I-FS-CBT, but the session organization was modified for a closed group format. The group treatment was designed to provide didactic presentation of coping skills and motivational enhancement material, and group discussion and rehearsal of new skills within a supportive atmosphere that facilitated mutual emotional support and support for abstinence. The first session of G-FS-CBT was 2 hours; remaining sessions were 90 minutes.

In-person follow-up interviews were done at 3, 9, and 15 months post-session 1.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* have a current (past year) Diagnostic and Statistical Manual-IV (DSM-IV) alcohol dependence diagnosis
* used alcohol in the 60 days prior to telephone screening

Exclusion Criteria:

* have psychotic symptoms in the past six months
* gross cognitive impairment
* current physiological dependence on any illicit drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants only
Enrollment: 155 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2014-04-28 (Actual); Study Completion 2014-04-28 (Actual)

PRIMARY OUTCOMES:
Percent Drinking Days (PDD) | Change from baseline across 15 months post-session 1
  Derived from Timeline Followback (TLFB)
Percent Heavy Drinking Days (PHDD) | Change from baseline across 15 months post-session 1
  Derived from TLFB; Defined as 4 or more standard drinks per day
Mean Drinks Per Drinking Day (MDPDD) | Change from baseline across 15 months post-session 1
  Derived from TLFB

SECONDARY OUTCOMES:
Beck Depression Inventory II | Baseline and through study completion, about 15 months
  self-report questionnaire assessing depression symptoms over the prior two weeks (scores range 0-63) and higher scores indicate greater depression symptomatology. All item scores are summed to attain a total score.
Anxiety | Baseline and through study completion, about 15 months
  Assessed anxiety symptoms in the last week (scores range 0-63) with higher scores indicating higher anxiety symptomatology. Item scores summed to attain total score.
Sociotropy-Autonomy Scale | Baseline and through study completion, about 15 months
  Measures the extent of an individual's concern with others' opinion of herself (sociotropy) and self-confidence, behavioral and emotional independence (autonomy). Sociotropy sub scale ranges from 0 to 64 with higher scores indicating higher sociotropy. Average Sociotropy Scores are attained by averaging items, with total scores from 0 to 4. Autonomy sub scale Score range from 0 to 44 with higher scores indicating greater autonomy. Average Autonomy Scores are attained by averaging items, with total scores from 0 to 4.
Coping Strategies Scale | Baseline and through study completion, about 15 months
  Assessed use frequency of 30 strategies to cope with alcohol use and non-alcohol related situations, on a scale of 1 (never) to 4 (frequently) for a mean score across all items
Situational Confidence Scale 8 | Baseline and through study completion, about 15 months
  Measured self-efficacy to abstain from alcohol use in high-risk situations; each item is rated 0% to 100% for a global confidence score.
Important People Inventory | Baseline and through study completion, about 15 months
  Assessed social network structure, network drinking, and network response to drinking and abstinence. Percentage of network accepting/encouraging abstinence and percentage of network abstainers/in recovery were used.
Self care | Baseline and through study completion, about 15 months
  Assessed 8 domains of self-care: seek medical care, have free time, pleasurable activities, social contact, attend treatment, exercise, do nice things for oneself, buy nice things for oneself
Inventory of Personal Problems | Baseline and through study completion, about 15 months
  Assessed problems in 10 interpersonal domains, rated on a 0 to 4 scale. A total sum score was used for this study; higher scores reflect more interpersonal problems
Group Environment Scale Form R | Baseline and through study completion, about 15 months
  Measured 10 group process subscales (e.g., Cohesiveness, Leader Support, Order/Organization, Expressiveness, Anger/Aggression), each with a mean scale score for 4 items rated on a 0-4 scale.

OTHER OUTCOMES:
End of Treatment Questionnaire | 3 months post session 1
  Measured client ratings of helpfulness of therapy elements on a 7 point scale of -3 (greatly harmful), -2, -1, 0 (neutral), +1, +2, +3 (greatly helpful).
Working Alliance Inventory - Short Form | Weekly during Treatment, about 15 weeks
  12-item self-report measure of the therapeutic alliance (7-point scale with a total possible score of 84)
Therapy Integrity Rating Scale | Weekly during treatment, about 15 weeks
  39 five-point Likert scale items to assess domains common to both treatment conditions (e.g., general interventions, female-specific interventions, common factors) and unique to a single treatment condition (e.g., group therapy interventions)
Therapist Checklist | Weekly during Treatment, about 15 weeks
  Coding treatment components delivered in each session from 3 to 0 as thoroughly, moderately, minimally, or not covered

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth E Epstein, PhD, Principal Investigator — Rutgers, The State University of New Jersey